CLINICAL TRIAL: NCT01216020
Title: Multiinstitutional Open Label Randomized Phase II Study Comparing Cetuximab and Radiotherapy Versus Cisplatin and Radiotherapy as Firstline Treatment for Patients With Locally Advanced Squamous Cell Carcinoma of the Head and Neck (LA-NHSCC)
Brief Title: Cetuximab Plus Radiotherapy Versus Cisplatin Plus Radiotherapy in Locally Advanced Head and Neck Cancer
Acronym: CTXMAB+RT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient recruitment
Sponsor: Azienda USL 4 Prato (Other)
Collaborators: Università degli Studi di Brescia (Other)
Responsible Party: Principal Investigator, STEFANO M. MAGRINI, PROF, PROF, Azienda USL 4 Prato
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: eudract 2010-021552-26
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Head and Neck Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Pharyngeal Neoplasms
Keywords: Head and Neck Cancer; Radiotherapy; Cetuximab; Cisplatin
MeSH Terms: conditions — Head and Neck Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Pharyngeal Neoplasms | interventions — Cetuximab; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cetuximab plus radiotherapy (Experimental): Cetuximab given one week before radiotherapy (loading dose, 400 mg/m2) plus weekly (250 mg/m2), concomitant with radiotherapy (7O Gy on clinically involved sites).
  Interventions: Drug: cetuximab
- cisplatin plus radiotherapy (Active Comparator): CDDP 40 mg/mq in a single weekly 1-hour infusion concomitant to radiotherapy: (70 Gy to clinically involved sites)
  Interventions: Drug: cisplatin (associated to radiotherapy)

INTERVENTIONS:
Drug: cetuximab — * Cetuximab is given according to the standard mode of administration: "loading dose" : 400 mg/m2 one week before the start of radiotherapy (week -1), followed by a weekly dose of 250 mg/m2 during the weeks of the treatment with radiotherapy.
  * Radiotherapy: Doses: Clinical sites of disease (T e N) : total dose of 70 Gy given with a fractional dose of 2 Gy/day; "prophylactic" nodal volume (N) : total dose of 50 Gy given with a fractional dose of 2 Gy/day ; Treatment technique: conformal 3D. Intensity modulated radiotherapy (IMRT), also with simultaneous boost (SIB), is allowed.
  Other Names: Erbitux
  Arms: cetuximab plus radiotherapy
Drug: cisplatin (associated to radiotherapy) — * CDDP dose: 40 mg/mq in a single weekly 1-hour infusion preceded by adequate hydration, diuretics e antiemetic premedication.
  * Radiotherapy: Doses: Clinical sites of disease (T e N) : total dose of 70 Gy given with a fractional dose of 2 Gy/day; "prophylactic" nodal volume (N) : total dose of 50 Gy given with a fractional dose of 2 Gy/day ; Treatment technique: conformal 3D. Intensity modulated radiotherapy (IMRT), also with simultaneous boost (SIB), is allowed.
  Other Names: Cisplatin
  Arms: cisplatin plus radiotherapy

SUMMARY:
BACKGROUND:

Concomitant radiotherapy and cisplatin (CDDP) based chemotherapy is the standard treatment for LA-NHSCC. This combined modality treatment is linked with considerable acute local and systemic toxicity.EGFR is overexpressed in 90-100% of the HNSCC cases and is considered an unfavourable prognostic marker. EGFR costitutive activation is linked with HNSCC pathogenesis.

Cetuximab is a monoclonal anti-EGFR antibody blocking the activation of the receptor and signal transduction. Cetuximab combined with radiotherapy is superior to radiotherapy only in the treatment of LA-HNSCC and is characterized by an acceptable toxicity profile.

RATIONALE:

A direct comparison between concomitant chemoradiotherapy with Cisplatin and the concomitant treatment with radiotherapy associated to cetuximab does not exist.

STUDY DESIGN:

Arm A: Radical radiotherapy (doses and volumes) concomitant with chemotherapy with Cisplatin (40 mg/mq/week) Arm B: Radical radiotherapy (doses and volumes) concomitant with therapy with the monoclonal antibody Cetuximab (400 mg/m2 ["loading dose"] and subsequently 250 mg /m2/week)

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

Evaluation and comparison of the compliance of the two treatments;

SECONDARY OBJECTIVES:

Evaluation and comparison of the grade and incidence of acute toxicity; Evaluation and comparison of local control; Evaluation and comparison of event free survival (both local control and distant metastases); Evaluation and comparison of cause specific and overall survival.

INCLUSION/EXCLUSION CRITERIA

* Histologically confirmed squamous cell carcinoma (biopsy obtained from the tumor and/or from its lymphnodal metastases) originating from oral cavity, oropharynx, hypopharinx, supraglottic larynx;
* Locally advanced disease, defined by one of the following criteria: every T, N+, M0 ( T1, N1 cases excluded); T3-4, N0, M0;
* Not a nasopharynx, paranasal sinuses, salivary glands tumor;
* General conditions and concomitant diseases not considered a contraindication for chemotherapy or curative radiotherapy;
* No other surgical, chemotherapeutic or radiotherapic treatments for ENT region tumors or for tumors of other anatomical sites (with the exception of non-melanoma cutaneous tumors and of the carcinoma in situ of the uterine cervix and of other solid tumors whose primary treatment has been completed more than 3 years before the accrual in this study and never relapsed since primary treatment (the patient having been since then continuously disease- free);
* Availability for follow-up;
* Signed informed consent;
* An interval of maximum 3 weeks between staging procedures for local disease and randomization
* An interval of maximum 2 weeks between randomization and the onset of the treatment

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed squamous cell carcinoma (with biopsy on the primary and / or lymph node metastases) of the oral cavity, oropharynx, hypopharynx, larynx supraglottix;
* Locally advanced disease, defined by one of the following criteria: any T, N +, M0 (excluding T1, N1), T3-4, N0, M0;
* Not cancer nasopharynx or paranasal sinuses or salivary glands;
* General conditions and associated diseases which does not allow to perform chemotherapy or radiotherapy in a radical view;
* No other surgical treatments, chemotherapy or radiotherapy for cancer of head and neck or elsewhere, except non-melanoma skin cancer or in situ cervical cancer and other solid tumors for which radical treatment has been completed > three years prior to enrollment in the study and for which the patient has remained continuously free of disease;
* Accessibility to follow-up;
* Signing of informed consent;
* Interval between examinations of local staging and randomization, maximum 3 weeks
* Interval between randomization and initiation of treatment, maximum 2 weeks

Exclusion Criteria:

* Age <18 years
* ECOG performance status > 0-1
* Hemoglobin <9 g / dL
* Counts of granulocytes, total <1.5 x 10 ^ 9 / L
* Platelet count <100 x 10 ^ 9 / L
* Bilirubin> 1.5 times upper limit of normal (ULN)
* AST or ALT> 3 times ULN
* Creatinine clearance > 50 mL/min
* Mg > 0.5 mmol/L
* Pregnancy or lactation
* Presence of allergy to study drug or to the excipients used in their formulation
* Peripheral neuropathy ≥ grade 2 (CTCAE v3.0)
* Hearing loss / tinnitus ≥ grade 3 (CTCAE v3.0)
* One of the following conditions:

  * Myocardial infarction within 12 months prior to randomization
  * Severe congestive heart failure
  * Unstable angina
  * Cardiomyopathy in act
  * Ventricular arrhythmia
  * uncontrolled hypertension
  * Severe psychotic disorders in act
  * Severe infection in act
  * Any other serious illness that could interfere with the administration of the therapy provided by the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2015-05-20 (Actual); Study Completion 2015-05-20 (Actual)

PRIMARY OUTCOMES:
Compliance | weekly during treatment
  Evaluation and comparison of the compliance of the two treatments arms

SECONDARY OUTCOMES:
event free survival | bimonthly for two years, every 6 months thereafter
  Evaluation and comparison of the event free survival (both local control and distant metastases)
acute toxicity | Weekly during treatment.
  Evaluation and comparison of the grade and incidence of acute toxicity.
Local control | bimonthly for two years after treatment, every six months thereafter
  Evaluation and comparison of local control
cause specific survival | bimonthly after treatment for two years, then every 6 months
  Evualation and comparison of cause specific survival
overall survival | bimonthly after treatment for two years, then every 6 months
  evaluation and comperison of overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Stefano M Magrini, Prof, Study Chair — Radiotherapy Dept., Brescia Hospital and Brescia University
Locations (7):
- Italy (7):
  - Radiotherapy Dept., Arezzo Hospital, Arezzo
  - Radiotherapy Dept., Brescia University and Medical Oncology Dept., Brescia Hospital, Brescia
  - Radiotherapy Dept., Florence University, Florence
  - Radiotherapy Dept., Genoa University, Genoa
  - Radiotherapy Dept., Azienda USL 4 Prato, Prato
  - Radiotherapy Dept., Siena University, Siena
  - Radiotherapy Dept., Turin University, Torino

REFERENCES:
- [Derived] Buglione M, Maddalo M, Corvo R, Pirtoli L, Paiar F, Lastrucci L, Stefanacci M, Belgioia L, Crociani M, Vecchio S, Bonomo P, Bertocci S, Borghetti P, Pasinetti N, Triggiani L, Costa L, Tonoli S, Grisanti S, Magrini SM. Subgroup Analysis According to Human Papillomavirus Status and Tumor Site of a Randomized Phase II Trial Comparing Cetuximab and Cisplatin Combined With Radiation Therapy for Locally Advanced Head and Neck Cancer. Int J Radiat Oncol Biol Phys. 2017 Mar 1;97(3):462-472. doi: 10.1016/j.ijrobp.2016.10.011. Epub 2016 Oct 20. PMID 27986347